CLINICAL TRIAL: NCT01795326
Title: Assessment of Physician Behavior Regarding Metabolic Monitoring of Patients Treated With SEROQUEL® (Quetiapine Fumarate) Tablets and SEROQUEL® (Quetiapine Fumarate) Extended Release Tablets in Selected Countries in the EU
Brief Title: Physician Survey on Monitoring of Patients Treated With Quetiapine
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1443C00127
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: Effectiveness of risk minimization; Metabolic monitoring; Seroquel®; Seroquel® XR/quetiapine fumarate
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Germany: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- United Kingdom: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Spain: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Hungary: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Netherlands: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Sweden: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Romania: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
- Italy: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.

SUMMARY:
A physician survey to document receipt of metabolic educational materials and assess behavior of physicians in following messages communicated through the educational materials

DETAILED DESCRIPTION:
Assessment of physician behavior regarding metabolic monitoring of patients treated with SEROQUEL® (quetiapine fumarate) Tablets and SEROQUEL® (quetiapine fumarate) Extended Release Tablets in selected countries in the EU

ELIGIBILITY:
Inclusion Criteria:

* Physicians targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.

Exclusion Criteria:

* Physicians who have participated in a survey involving SEROQUEL® / SEROQUEL® XR in the past six months are not eligible to participate in this survey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A sample of physicians who were targeted to receive the metabolic educational materials and either currently prescribe or have the potential to prescribe SEROQUEL® or SEROQUEL® XR.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determination via survey whether physicians or someone in their practice perform monitoring of patients treated with Seroquel or Seroquel XR for metabolic issues related to treatment; refer their patients to another physician for monitoring. | Over 6- 8 weeks.
Determination via survey whether physicians monitor tests for hyperlipidemia in patients who are taking Seroquel or Seroquel XR. | Over 6- 8 weeks.
Determination via survey whether physicians monitor for signs and symptoms of hyperglycemia in patients who are taking Seroquel or Seroquel XR. | Over 6- 8 weeks.
Determination via survey whether physicians monitor blood glucose in patients with diabetes or monitor patients with risk factors for diabetes for worsening of glycemic control if they are taking Seroquel or Seroquel XR. | Over 6- 8 weeks.
Determination via survey whether physicians monitor weight at initiation of treatment with Seroquel or Seoquel XR and on a regular basis after initiating treatment. | Over 6- 8 weeks.

SECONDARY OUTCOMES:
Determination via survey whether physicians counsel patients taking with Seroquel or Seroquel XR on healthy eating, exercise, and healthy lifestyle improvements. | Over 6- 8 weeks.
Determination via survey whether physicians received educational information relevant to the issues in the survey from AstraZeneca. | Over 6- 8 weeks.
Determination via survey whether physicians read the educational information. | Over 6- 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brody, MPH, Principal Investigator — AZ